CLINICAL TRIAL: NCT06028152
Title: Adapting an Advance Care Planning Intervention and Delivery Model for Use With Patients With Cancer and Their Caregivers
Brief Title: Using an End-of-life Conversation Game to Engage Patients With Cancer in Advance Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Van Scoy, Professor of Medicine, Humanities and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023029
Record Dates: First submitted 2023-08-29; First posted 2023-09-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Lung Cancer; Genito Urinary Cancer
Keywords: Advance Care Planning; Advance Directives; Terminal Illness
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Game participants (Experimental): All participants will engage in playing the end-of-life conversation game called "Hello", which involves answering open-ended questions about medical decision making and end-of-life issues.
  Interventions: Other: End-of-life conversation game called "Hello"

INTERVENTIONS:
Other: End-of-life conversation game called "Hello" — To play 'Hello', players are provided 32 open-ended questions in a prearranged order and an equal number of game chips. A player reads aloud the first question. Players then individually write down their answers, and take turns sharing answers with the group (players can opt to pass). Players control how long they share, what they share, and when they are ready to proceed to the next question. During the conversation, players may choose to acknowledge others for a particularly thoughtful, poignant, or even funny comment by giving them a chip. A simple pre-game coin flip determines whether the player with the most chips 'wins' the game ('heads'), or the player with the least amount of chips wins the game ('tails').
  Other Name: Previously named "My Gift of Grace"

SUMMARY:
The goal of this clinical trial is to explore feasibility, acceptability, and effectiveness of end-of-life conversation game "Hello" as a tool to help individuals with breast, lung, and/or genito-urinary cancers treated at Penn State Cancer Institute and their loved ones perform advance care planning. The main questions it aims to answer are:

* What modifications and/or adaptations are necessary to Hello for use in cancer populations?
* How do different delivery models compare for recruitment in terms of feasibility and efficiency?

Participants will:

* Complete pre-game questionnaires
* Play the Hello game
* Complete post-game questionnaires
* Participate in a focus group

DETAILED DESCRIPTION:
Previous studies conducted by the investigators have shown that the Hello game demonstrates successful ACP engagement in general populations, but has yet to be tailored to meet the unique needs of patients with advanced cancer and their caregivers. Outlining their care preferences by engaging in ACP is an important aspect of care according to patients with advanced cancer. However, only 55% of patients with advanced cancer patients have participated in ACP. These patients have substantial bio-psycho-social stressors that distinguish their ACP needs from others. Tailoring established interventions that foster high quality conversations about medical treatment preferences and end-of-life issues (such as the Hello game) is critically important for this population given its unique needs. As evidenced by qualitative interviews with >200 participants, the Hello game creates a safe environment for sensitive conversations about end-of-life issues and inspired sharing of rich perspectives, with no reported adverse events, excessive burden, or negative emotional effects. That said, the intervention must be adapted for patients with cancer, particularly those with advanced cancer and their caregivers.

Additionally, while several effective ACP interventions exist (including Hello), how best to disseminate these interventions has not been rigorously or systematically studied. In other ongoing and previous studies, the investigators have demonstrated success in both engaging individuals living in underrepresented communities in ACP and successfully enrolling them in interventional research about ACP. The investigators credit these successes to their unique intervention delivery approach called the Community Based Delivery Model (CBDM). The CBDM overcomes key barriers to ACP (such as healthcare distrust, resistance, and hesitancy to discuss end-of-life issues) by leveraging established community connections to recruit participants to participate in ACP interventions as well as research. In the CBDM, trusted community "hosts" (who are leaders from local hospice organizations, senior centers, health agencies) invite participants to attend an ACP event. They introduce the research team to the attendees who may choose to participate in the ACP activity, the research, or both. Hosts are provided with marketing materials and utilize their community network channels to advertise the event. This model allows for research to be conducted more easily within hard to reach and underserved communities such as Black, Hispanic and rural communities- much like the most remote communities across the PSCI's 28-county catchment area.

Patients with cancer, however, are unique, and may require an alternative approach that involves partnering with their oncology care team to introduce the concept of ACP and encourage participation in ACP and research. Notably, there is evidence that patients are more likely to engage in ACP when recommended by their physician, so how best to approach ACP for cancer patients is unknown. A common approach to ACP intervention research is to use a Healthcare Based Delivery Model (HBDM). In contrast to the CBDM, the HBDM is positioned within the healthcare system (i.e., clinic-based recruitment) as the ACP intervention is recommended by the patient's clinician (rather than through community-based outreach groups). For this intervention delivery approach, research assistants support interactions between clinicians (providers or nurses) to find appropriate patients and garner interest in performing ACP. This model is commonly used to recruit patients for clinical trials, including ACP interventions. For patients with cancer, the HBDM may have some advantages over the CBDM, given the close bonds that form between a patient and clinical care team as they interact frequently during active treatments such as infusions and radiation that often span several hours and weeks. Leveraging these therapeutic relationships may support greater acceptance of opportunities to broach ACP than a community-based model, but this remains unknown.

ELIGIBILITY:
Inclusion Criteria Cancer Patient:

* Adults (> 18 years old)
* Able to speak and read English
* Be an individual diagnosed with breast, lung, or genitourinary/prostate cancer as verified by primary oncologist or is the chosen caregiver for a participant with those cancers
* Receives care at Penn State Health or is the chosen caregiver for a participant treated at Penn State Health

Inclusion Criteria Caregiver/Loved one:

* Adults (> 18 years old)
* Able to speak and read English and/or Spanish
* Be the chosen caregiver for a participant with cancer

Exclusion Criteria Cancer Patient:

* Anyone <18 years of age
* Anyone unable to speak and read English
* Unable to provide informed consent
* Receives cancer care exclusively outside of Penn State Health

Exclusion Criteria Caregiver/Loved one:

* Anyone <18 years of age
* Anyone unable to speak and read English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Experiences and perceptions of intervention | Immediately post-intervention
  Group discussions held with patients with cancer and their caregivers to collect qualitative data on acceptability of the game, necessary modifications for use in patients with cancer and their caregivers, and other feedback and opinions on the game experience.

SECONDARY OUTCOMES:
Advance Care Planning Engagement Measure | Baseline
  This 4-item short-version survey measures readiness to perform ACP.
Advance Care Planning Surrogate Decision Maker Engagement Measure | Baseline
  This 17-item survey measures surrogate decision maker readiness to perform ACP.
Satisfaction of Intervention Measure | Immediately post-intervention
  This 8-item survey measures participants' satisfaction with the conversation. Each item is scored on a 1-7 scale with 1 being lowest conversation satisfaction. The items are averaged for the final score ranging 1-7 with 7 indicating the highest conversation satisfaction.
Acceptability of Intervention Measure | Immediately post-intervention
  This 3-item survey measures participants' perceived acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Van Scoy, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimbel K, Hayes M, Bucher M, Calo WA, Garg T, Joshi M, Kuntz H, Murphy TE, VanDyke E, Wasserman E, Van Scoy LJ. Facilitating Advance Care Planning Conversations Among Patients With Cancer and Their Care Partners Utilizing a Conversation Game: A Pilot Study. Cancer Rep (Hoboken). 2025 Jun;8(6):e70250. doi: 10.1002/cnr2.70250. PMID 40528532